CLINICAL TRIAL: NCT02302430
Title: Psychobiological Assessment and Enhancement of Team Cohesion and Psychological Resilience Using a Virtual Team Cohesion Test.
Brief Title: Intranasal Oxytocin and Enhancement of Team Cohesion
Acronym: ECHO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joshua Woolley, Principal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 14-15259
Record Dates: First submitted 2014-11-14; First posted 2014-11-27 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Unit Cohesion
Keywords: Cohesion; Oxytocin; Trust; Virtual-reality
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: SOLO arm and ECHO arm -- Acquainted, Unacquainted
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Treatment group will receive either 20IU or 40IU intranasal oxytocin
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo group will receive a saline nasal spray
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Drug: Oxytocin — 20 International Units Intranasal Oxytocin
  Other Names: Syntocinon
  Arms: Treatment
Other: Placebo comparator — Saline nasal spray
  Arms: Placebo

SUMMARY:
This study attempts to identify the psychological, behavioral, physiological, and hormonal predictors and mechanisms of an individual's ability to develop cohesion in a group working together as a team; and examine if administration of the prosocial neuropeptide oxytocin enhances the development of team cohesion. Through a deeper understanding of the underlying psychobiological predictors and mechanisms of team cohesion, the prospective identification of individuals whose unique characteristics promote or inhibit the development of group cohesion will become possible.

DETAILED DESCRIPTION:
The investigators will study up to one thousand subjects who will be randomized into same-gendered teams of three or volunteer as acquainted groups of three . Teams will be randomized to receive oxytocin or placebo. The investigators will first measure baseline personality traits including prosocial orientation. Cohesion will then be measured using a cooperative, virtual unmanned aerial vehicle (UAV) flying mission. All online behavior will be recorded within the task and all offline, real world, behavior will be video recorded throughout the study by digital cameras for later behavioral coding. To measure biobehavioral synchrony, autonomic physiology will be recorded and saliva samples will be taken throughout behavioral testing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-28
* Speak English
* Ability to use a nasal spray

Exclusion Criteria:

* Positive urine pregnancy test
* History of psychiatric or neurologic disorder
* Use of illicit drugs in the past month
* History of moderate-severe alcohol use disorder as defined by DSM-V criteria
* Sensitivity to preservatives (in particular E 216, E 218 and chlorobutanol hemihydrate)
* Nasal obstruction, discharge, or bleeding
* Habitually drinks large volumes of water
* Taking testosterone, estrogen/progesterone supplement, or serotonin-1a receptor agonists/antagonists
* Currently meets Diagnostic and Statistical Manual-5 (DSM-V) criteria for severe major depressive disorder with suicidal thoughts or actions

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 486 (Actual)
Dates: Start 2015-10; Primary Completion 2018-05 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change in score on computer game task | Baseline, 2 hours after drug/placebo administration
  Subjects will work together in groups of 2-4 performing a computer-based task flying a virtual plane.

SECONDARY OUTCOMES:
Change is psychophysiological output | Time based variability analyzed for 5 minute or 20 minute events
  Cardiac measures (HRV, Impedance) collected during computer based and group activities

CONTACTS AND LOCATIONS:
Overall Officials: Josh D Woolley, MD/PhD, Principal Investigator — University of California San Francisco, San Francisco Veterans Affairs Medical Center
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States